CLINICAL TRIAL: NCT06293677
Title: Upwards Initial Adjustment of Wide-Spectrum Antibiotic Dosage in Pediatric Oncology Patients With Febrile Neutropenia and Suspected Augmented Renal Clearance: A Randomized Controlled Trial With Therapeutic Drug Monitoring
Brief Title: Adjustment of Antibiotic Dosage in Pediatric Oncology Patients With Febrile Neutropenia and Augmented Renal Clearance
Acronym: DAR-ARC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Unisanté Centre universitaire de médecine générale et santé publique (Unknown); FORCE Fondation Recherche sur le Cancer de l'Enfant (Unknown)
Responsible Party: Principal Investigator, Pierre Alex Crisinel, Head of the Unit of Pediatric Infectious Diseases and Vaccinology, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01013
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Febrile Neutropenia
Keywords: Febrile neutropenia; Augmented Renal Clearance; Pediatric cancer; Therapeutic Drug monitoring TDM; Children; Wilde-spectrum antibiotic dosage; Glomerular filtration rate GFR
MeSH Terms: conditions — Febrile Neutropenia; Neoplasms | interventions — Meropenem

STUDY DESIGN:
Intervention Model Description: Our study is an open-label, re-randomized controlled trial in multi-episodes settings. So the care team, researchers and patients will be informed of the allocation group. Patients will be able to participate in each episode of febrile neutropenia. At each inclusion the patient may be in a different group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group 1c (Active Comparator): Group 1c includes patients with augmented renal clearance (ARC) who have been randomized to receive a standard dosage of antibiotic (méropenem or piperacilline-tazobactam)
  Interventions: Drug: Standard dosages of piperacillin-tazobactam or meropenem
- Intervention DAR-ARC Group 1i (Experimental): Group 1i (DAR-ARC) includes patients with ARC who have been randomized to receive an experimental dosage of antibiotic (méropenem or piperacilline-tazobactam)
  Interventions: Drug: Dosage Adjustment Rules for Augmented Renal Clearance (DAR-ARC) for piperacillin-tazobactam and meropenem
- Control Group 2 (Active Comparator): Control Group 2 includes patients with normal or decreased renal function who will receive standard dosage of antibiotic (méropenem or piperacilline-tazobactam)
  Interventions: Drug: Standard dosages of piperacillin-tazobactam or meropenem

INTERVENTIONS:
Drug: Dosage Adjustment Rules for Augmented Renal Clearance (DAR-ARC) for piperacillin-tazobactam and meropenem — Meropenem dosages according to eGFR [mL/min/1.73 m²] :
  eGFR 120-149 : 40 mg/kg q6 h eGFR 150-199 : 30 mg/kg q4h eGFR 200-299 : 40 mg/kg q4h eGFR >/= 300 : 40 mg/kg q4h
  Piperacillin-tazobatam dosages according to eGFR [mL/min/1.73 m²] :
  eGFR 120-149 : 150 mg/kg q6 h eGFR 150-199 : 120 mg/kg q4h eGFR 200-299 : 150 mg/kg q4h eGFR >/= 300 : 180 mg/kg q4h
  The maximum doses for the antibiotic prescription before the first drug monitoring will be 2gr of MER every 4 hours and 4gr of PIP every 4 hours.
  The duration of infusion will be set to 2 h.
  Arms: Intervention DAR-ARC Group 1i
Drug: Standard dosages of piperacillin-tazobactam or meropenem — Meropenem dosages according to eGFR [mL/min/1.73 m²] :
  eGFR> 50 : 40mg/kg q8h eGFR 25-49 : 40mg/kg q12h eGFR 15-24 : 20mg/kg q12h
  Piperacillin-tazobactam :
  eGFR >50 : 100mg/kg q6h eGFR 20-49 : 50mg/kg q6h eGFR 15-29 : 50 mg/kg q8h
  Arms: Control Group 1c; Control Group 2

SUMMARY:
This clinical trial focuses on children with cancer who face infections after receiving chemotherapy. Chemotherapy affects the bone marrow, leading to a decrease in the production of certain white blood cells, particularly those that defend against bacterial infections (neutrophils). One significant concern is febrile neutropenia, where children experience a fever during a period of low white blood cell count. This condition often results from bacterial infections, necessitating prompt wide-spectrum antibiotic treatment. However, some children eliminate antibiotics in the urine too quickly during febrile neutropenia. Their kidneys function more than they normally do (renal hyperfiltration). This can lead to insufficient exposure to antibiotics to control the infection. The current standard antibiotic regimens do not account for this variable elimination rate. In this study we focus on two antibiotics used in this context: piperacillin-tazobactam and meropenem.

The main questions this study aims to answer are, in these children:

* Would higher doses of antibiotics result in better blood levels of antibiotics?
* Would they have more sides effects with higher antibiotics dosages?
* Would they recover more quickly with higher antibiotic doses? All patients will undergo a blood test upon hospital arrival, including an assessment of renal function. If renal function is normal or diminished, the patient will receive the standard antibiotic dose. Children with increased renal function will be randomly assigned to two groups during each episode of febrile neutropenia. One group will receive standard antibiotic dosages, while the other will receive higher doses to compensate for renal hyperfiltration. Throughout the study, antibiotic levels in the blood will be monitored for all patients. This monitoring will determine if target concentrations can be achieved more quickly with experimental dosages and will allow doctors to readjust the doses if needed.

DETAILED DESCRIPTION:
Background and Rationale In pediatric cancer patients, Augmented Renal Clearance (ARC) is a common factor that affects outcomes. Febrile neutropenia, a frequent occurrence during cancer treatment, requires anti-infective drugs for treatment. However, ARC increases the elimination of these drugs through glomerular filtration, posing a risk of antibiotics insufficient blood levels. This may lead to difficulties in managing infections and the risk of antibiotic-resistant bacterial strains emerging. Febrile neutropenia is often associated with ARC, and in these patients standard antibiotic dosages frequently miss target concentrations. We propose defining categories of renal hyperfiltration to adjust antibiotic dosages upward in pediatric patients with ARC.

To estimate renal function, molecules such as creatinine or cystatin C are routinely measured in the blood. Clinicians commonly rely on the Schwartz formula for determining the patients glomerular filtration rate (GFR) when adjusting antibiotic treatment. Although other formulas based on creatinine and/or cystatin C have been developed, their effectiveness in oncological patients with ARC remains unexplored. If these alternative formulas prove more effective in ARC situations, it may prompt a reconsideration of how we determine GFR in hyperfiltrating children.

Measurement and procedures Clinicians will decide if prescribe piperacillin-tazobactam or meropenem, according to the clinical situation. The trial will have 3 arms, the two control arms will receive standard dosages of antibiotics (non-hyperfiltrating patients, control group 2, and hyperfiltrating patients randomized to control group 1c). The third group, hyperfiltrating patients randomized to intervention group 1i, will receive experimental doses. The randomization will be made using REDCap®.

A TDM at trough level (Ctrough) of meropenem (MER) or piperacillin-tazobactam (PIP) will be systematically performed just before the fourth dose, and again before the fourth dose after each further dosage adaptation. The dosage will be adjusted if blood levels are outside the target therapeutic ranges. TDM will be monitored at least twice a week and more frequently in case of unfavorable clinical outcome or significant change in serum creatinine.

Objectives

Primary objective:

To compare the proportion of early achievement of antibiotic concentration targets in hyperfiltrating patients, using either standard dosage recommendations (control group, 1C) or a new set of Dosage Adjustment Rules for Augmented Renal Clearance (DAR-ARC) (intervention group, 1i).

Secondary objectives:

1. To compare the proportion of early achievement of antibiotic concentration targets (for MER or PIP) between non hyperfiltrating patients (control group 2) and the intervention group (1i).
2. To compare the mean/median duration of fever episodes between control groups and intervention group (1i)
3. To compare the incidence of intervention-drug adverse effects (CTCAE v5, grade 3 or higher, grade 2 judged to be probably/definitely related to study intervention and SAE) between the control groups (group 1c and 2) and the intervention group (1i)
4. To compare the proportion of patients requiring TDM-based readjustment of antibiotic dosages due to blood level below or above the target ranges between the control group 1c and the intervention group 1i, at any time during the antibiotic treatment.
5. To compare the eGFR estimated by creatinine-based Schwartz formula in comparison to creatinine and cystatin C based Schwartz formula, creatinine-based quadratic formula, combined creatinine and cystatin C Quadratic formulas, Zappitelli formula, and Schwartz-Lyon formula.

Statistical Considerations The proportion of achievement of the target ranges before the fourth antibiotic dose will be compared between the two randomized groups with a mixed effects logistic regression.

Duration of fever will be analyzed by the Kaplan-Meier method. Cox regression analysis will be used to evaluate if the intervention decreases duration of fever.

The occurrence of adverse events and the outcome of the febrile neutropenia episode will be compared between groups using a Chi-square test.

The use of TDM for further adjustment of MER and PIP dosage will be explored with descriptive statistics. A population pharmacokinetic description of MER and PIP concentration will be attempted.

To evaluate different eGFR formulas, we will calculate the mean difference in eGFR estimation for each formula compared to the creatinine-based Schwartz formula and determine a 95% confidence interval for each formula. Comparison between hyperfiltrating non hyperfiltrating will be made using student T-test or Kruskal-Wallis tests.

Unless otherwise stated, the α risk p -values reported will be two-sided and the nominal limit will be set to 0.05.

Risk / Benefit Assessment The risk of this study is over exposure to wide-spectrum antibiotics. This implies drugs dose-dependent adverse events.

High blood trough concentrations (Ctrough) of broad-spectrum antibiotics have been associated with reversible neurological and nephrological side effects in adults. The threshold level chosen in this protocol is well below the values for which there is a risk of a 50% increase in side effects for both antibiotics. Doses of MER and PIP excess of authorized doses, guided by therapeutic drug monitoring, have not been associated with additional toxicities in adults. The evaluation of renal clearance before the choice of dosage, daily clinical and biological monitoring and regular monitoring of Ctrough will limit risks.

The expected benefit will be improved circulating exposure to broad-spectrum antibiotics. This could allow better control of the infection with a more rapid and favorable clinical course.

ELIGIBILITY:
Patients' inclusion criteria

* Oncologic patients aged 2 months to 17 years (older than 60 days and younger than 18 years),
* High probability of febrile neutropenia during the study period
* Written informed consent from parents and adolescents older than 14 years

Patients' exclusion criteria

* Neutropenia not related to cancer and/or chemotherapy
* Refusal to participate
* Non-French speaking parents/patients older than 11 years old
* Absence of febrile neutropenia or agranulocytosis during the study period (secondary exclusion)

Febrile neutropenia episodes inclusion criteria

* Febrile neutropenia or agranulocytosis defined as:

  * Neutropenia: absolute neutrophils <500 cells/µL or agranulocytosis: absolute neutrophils <100 cells/µL or patients expected to be neutropenic in the next 24 hours due to ongoing chemotherapy
  * body temperature (tympanic or axillary) ≥38°C during at least one hour or a single T ≥38.5°C
* At least 2 weeks after the end of the previous antibiotic treatment for another included episode of febrile neutropenia.

Febrile neutropenia episodes exclusion criteria:

* Severe renal failure (GFR<15 mL/min/1.73 m²)
* Pregnancy
* Inability to obtain the first therapeutic drug monitoring (TDM) result within 72 hours of sampling (e.g. admission before or during public holidays laboratory closure)

Ages: 61 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Achievement of antibiotic concentration targets in the intervention group (1i) vs control groupe (1c) | During the first 24 hours of the intervention, before the fourth dose of antibiotic
  Intervention-drug blood concentration both above the lower limit and below the upper limit of the therapeutic target ranges on the first trough dosage before the fourth dose after treatment initiation.

SECONDARY OUTCOMES:
Achievement of antibiotic concentration targets in control group 2 | During the first 24 hours of the intervention, before the fourth dose of antibiotic
  Intervention-drug blood concentration both above the lower limit and below the upper limit of the therapeutic target ranges on the first trough dosage before the fourth dose after treatment initiation in group 2
Fever duration | During the intervention
  Duration of fever (T ≥38°C) after initiation of antibiotherapy (time between first dose of antibiotic and last measurement of T ≥38°C followed by at least 24 hours of T <38°C)
Side effects of antibiotic therapy | During the intervention and up to 2 weeks after
  Any relevant adverse event judged to be probably/definitely related to study intervention and all serious adverse events (SAEs)
Number of dosage adjustments required to achieve the target concentration | During the intervention
  Readjustment of the intervention drug dosage because of blood concentration either below the lower limit or above the upper limit of the therapeutic target ranges (at any time)
Difference between eGFR measured by creatinine-based Schwartz formula and other eGFR calculation formulas | Baseline, pre-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alex Crisinel, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitelier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersson J, Giske CG, Eliasson E. Standard dosing of piperacillin and meropenem fail to achieve adequate plasma concentrations in ICU patients. Acta Anaesthesiol Scand. 2016 Nov;60(10):1425-1436. doi: 10.1111/aas.12808. Epub 2016 Sep 21. PMID 27655029
- [Background] Scharf C, Paal M, Schroeder I, Vogeser M, Draenert R, Irlbeck M, Zoller M, Liebchen U. Therapeutic Drug Monitoring of Meropenem and Piperacillin in Critical Illness-Experience and Recommendations from One Year in Routine Clinical Practice. Antibiotics (Basel). 2020 Mar 21;9(3):131. doi: 10.3390/antibiotics9030131. PMID 32245195
- [Background] Udy AA, Roberts JA, Lipman J. Implications of augmented renal clearance in critically ill patients. Nat Rev Nephrol. 2011 Jul 19;7(9):539-43. doi: 10.1038/nrneph.2011.92. PMID 21769107
- [Background] Hirai K, Ihara S, Kinae A, Ikegaya K, Suzuki M, Hirano K, Itoh K. Augmented Renal Clearance in Pediatric Patients With Febrile Neutropenia Associated With Vancomycin Clearance. Ther Drug Monit. 2016 Jun;38(3):393-7. doi: 10.1097/FTD.0000000000000270. PMID 27172381
- [Background] Imani S, Buscher H, Marriott D, Gentili S, Sandaradura I. Too much of a good thing: a retrospective study of beta-lactam concentration-toxicity relationships. J Antimicrob Chemother. 2017 Oct 1;72(10):2891-2897. doi: 10.1093/jac/dkx209. PMID 29091190
- [Background] McDonald C, Cotta MO, Little PJ, McWhinney B, Ungerer JP, Lipman J, Roberts JA. Is high-dose beta-lactam therapy associated with excessive drug toxicity in critically ill patients? Minerva Anestesiol. 2016 Sep;82(9):957-65. Epub 2016 Apr 7. PMID 27054905
- [Background] de With K, Allerberger F, Amann S, Apfalter P, Brodt HR, Eckmanns T, Fellhauer M, Geiss HK, Janata O, Krause R, Lemmen S, Meyer E, Mittermayer H, Porsche U, Presterl E, Reuter S, Sinha B, Strauss R, Wechsler-Fordos A, Wenisch C, Kern WV. Strategies to enhance rational use of antibiotics in hospital: a guideline by the German Society for Infectious Diseases. Infection. 2016 Jun;44(3):395-439. doi: 10.1007/s15010-016-0885-z. PMID 27066980
- [Background] Andre P, Diezi L, Dao K, Crisinel PA, Rothuizen LE, Chtioui H, Decosterd LA, Diezi M, Asner S, Buclin T. Ensuring Sufficient Trough Plasma Concentrations for Broad-Spectrum Beta-Lactam Antibiotics in Children With Malignancies: Beware of Augmented Renal Clearance! Front Pediatr. 2022 Jan 5;9:768438. doi: 10.3389/fped.2021.768438. eCollection 2021. PMID 35083184